CLINICAL TRIAL: NCT03135262
Title: A Phase Ib/II Study Evaluating the Safety and Efficacy of Obinutuzumab in Combination With Idasanutlin and Venetoclax in Patients With Relapsed or Refractory Follicular Lymphoma and Obinutuzumab or Rituximab in Combination With Idasanutlin and Venetoclax in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Obinutuzumab in Combination With Idasanutlin and Venetoclax in Participants With Relapsed or Refractory (R/R) Follicular Lymphoma (FL) or Rituximab in Combination With Idasanutlin and Venetoclax in Participants With R/R Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision to terminate the study after Phase 1; will not proceed with Phase 2.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH39147; 2016-002480-34 (EudraCT Number)
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Follicular Lymphoma; Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse | interventions — RG7388; obinutuzumab; venetoclax; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose-Escalation Cohort: FL (Experimental): Induction Treatment: Participants will receive either Regimen A or Regimen B. Regimen A: Participants will receive either obinutuzumab on Days 1, 8, 15 of Cycle 1 and then on Day 1 of Cycles 2 to 6; idasanutlin and venetoclax on Days 1 to 5 of Cycles 1 to 6 or obinutuzumab on Days 1, 8, 15 on Cycle 1 and then on Day 1 of Cycles 2 to 6; idasanutlin on Days 1 to 5 and venetoclax on Days 1 to 10 of Cycles 1 to 6. Regimen B (in bridging cohort): Participants will receive obinutuzumab alone in Cycle 1 and obinutuzumab with idasanutlin and venetoclax (both at maximum tolerated dose [MTD] established from Regimen A) in Cycles 2 to 6. Post-Induction Treatment (Maintenance Treatment): Participants will receive obinutuzumab every 2 months for 24 months; idasanutlin and venetoclax for 6 months.
  Interventions: Drug: Idasanutlin; Drug: Obinutuzumab; Drug: Venetoclax
- Dose-Escalation Cohort: DLBCL (Experimental): Induction Treatment: Participants will receive either obinutuzumab on Days 1, 8, 15 of Cycle 1 and then on Day 1 of Cycles 2 to 6; idasanutlin and venetoclax on Days 1 to 5 of Cycles 1 to 6 or obinutuzumab on Days 1, 8, 15 on Cycle 1 and then on Day 1 of Cycles 2 to 6; idasanutlin on Days 1 to 5 and venetoclax on Days 1 to 10 of Cycles 1 to 6. In bridging cohort, participants will receive rituximab on Day 1 of Cycles 1 to 6 and idasanutlin and venetoclax (both at MTD) in Cycles 1 to 6. Post-Induction Treatment (Consolidation Treatment): Participants will receive obinutuzumab or rituximab (according to study treatment received in the induction) every 2 months for 6 months; idasanutlin and venetoclax for 6 months.
  Interventions: Drug: Idasanutlin; Drug: Obinutuzumab; Drug: Venetoclax; Drug: Rituximab
- Expansion Cohort: FL (Experimental): Induction Treatment: Participants will receive idasanutlin and venetoclax at the RP2D of the selected regimen (Regimen A or B) identified during the dose-escalation phase in combination with obinutuzumab. Regimen A: Participants will receive either obinutuzumab on Days 1, 8, 15 of Cycle 1 and then on Day 1 of Cycles 2 to 6; idasanutlin and venetoclax on Days 1 to 5 of Cycles 1 to 6 or obinutuzumab on Days 1, 8, 15 on Cycle 1 and then on Day 1 of Cycles 2 to 6; idasanutlin on Days 1 to 5 and venetoclax on Days 1 to 10 of Cycles 1 to 6. Regimen B (in bridging cohort): Participants will receive obinutuzumab alone in Cycle 1 and obinutuzumab with idasanutlin and venetoclax in Cycles 2 to 6. Post-Induction Treatment (Maintenance Treatment): Participants will receive obinutuzumab every 2 months for 24 months; idasanutlin and venetoclax for 6 months.
  Interventions: Drug: Idasanutlin; Drug: Obinutuzumab; Drug: Venetoclax
- Expansion Cohort: DLBCL (Experimental): Induction Treatment: Participants will receive rituximab on Day 1 of Cycles 1 to 6; idasanutlin and venetoclax (both at RP2D) on Days 1 to 5 of Cycles 1 to 6 or rituximab on Day 1 of Cycles 1 to 6; idasanutlin on Days 1 to 5 and venetoclax on Days 1 to 10 of Cycles 1 to 6. Post-Induction Treatment (Consolidation Treatment): Participants will receive rituximab every 2 months for 6 months; idasanutlin and venetoclax for 6 months.
  Interventions: Drug: Idasanutlin; Drug: Venetoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Idasanutlin — Induction Treatment: Idasanutlin tablets will be administered orally once daily at escalated doses (starting dose 100 milligrams [mg], maximum 600 mg). Post-Induction Treatment: The dose and regimen will be determined by the Sponsor after review of all relevant data. The dose for maintenance/consolidation will not exceed the dose the participant received during induction.
Drug: Obinutuzumab — Participants will receive a fixed dose of obinutuzumab, 1000 mg by intravenous (IV) infusion on Days 1, 8 and 15 of Cycle 1 and on Day 1 of each subsequent cycle (Cycles 2 to 6) (each cycle = 28 days) during induction treatment, and on Day 1 of every other month during maintenance treatment (eligible participants with FL only) or during consolidation treatment (eligible participants with DLBCL only).
  Arms: Dose-Escalation Cohort: DLBCL; Dose-Escalation Cohort: FL; Expansion Cohort: FL
Drug: Venetoclax — Induction Treatment: Venetoclax tablets will be administered orally once daily at escalated doses (starting dose 200 mg, maximum 800 mg). Post-Induction Treatment: The dose and regimen will be determined by the Sponsor after review of all relevant data. The dose for maintenance/consolidation will not exceed the dose the participant received during induction.
Drug: Rituximab — Rituximab will be administered by IV infusion at a dose of 375 milligrams per square meter (mg/m^2) on Day 1 of Cycles 1-6 during induction treatment and on Day 1 of every other month during consolidation treatment.
  Arms: Dose-Escalation Cohort: DLBCL; Expansion Cohort: DLBCL

SUMMARY:
This Phase Ib/II, open-label, multicenter, non-randomized, dose-escalation study will evaluate the safety, efficacy, and pharmacokinetics of obinutuzumab in combination with idasanutlin and venetoclax in participants with R/R FL and obinutuzumab or rituximab in combination with idasanutlin and venetoclax in participants with R/R DLBCL. The study will include an initial dose-escalation phase followed by an expansion phase. The dose-escalation phase is designed to determine the recommended phase II doses (RP2Ds) and regimen for idasanutlin and venetoclax in combination with obinutuzumab for FL participants and in combination with rituximab for DLBCL participants.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* B-cell lymphoma classified as either of the following: R/R FL after treatment with at least one prior chemoimmunotherapy regimen that included an anti-cluster of differentiation 20 (CD20) monoclonal antibody; R/R DLBCL after treatment with at least one prior chemoimmunotherapy regimen that included an anti-CD20 monoclonal antibody in participants who are not eligible for second line combination chemotherapy and autologous stem-cell transplantation, have failed second line combination chemotherapy, or experienced disease progression following autologous stem-cell transplantation
* Histologically documented CD20-positive lymphoma
* Fluorodeoxyglucose (FDG)-avid lymphoma (that is [i.e.], PET-positive lymphoma)
* At least one bi-dimensionally measurable lesion (greater than [>] 1.5 centimeters [cm] in its largest dimension by CT scan or magnetic resonance imaging [MRI])
* Availability of a representative tumor specimen and the corresponding pathology report for retrospective central confirmation of the diagnosis of FL or DLBCL

Exclusion Criteria:

* Known CD20-negative status at relapse or progression
* Prior allogeneic stem-cell transplantation (SCT)
* Completion of autologous SCT within 100 days prior to Day 1 of Cycle 1
* Prior standard or investigational anti-cancer therapy as specified: Radioimmunoconjugate within 12 weeks prior to Day 1 of Cycle 1; Monoclonal antibody or antibody-drug conjugate within 4 weeks prior to Day 1 of Cycle 1; Radiotherapy, chemotherapy, hormonal therapy, or targeted small-molecule therapy within 2 weeks prior to Day 1 of Cycle 1
* Clinically significant toxicity (other than alopecia) from prior therapy that has not resolved to Grade less than or equal to (</=) 2 (according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.0) prior to Day 1 of Cycle 1
* Grade 3b FL
* History of transformation of indolent disease to DLBCL (expansion-phase only)
* Central nervous system lymphoma or leptomeningeal infiltration
* Treatment with systemic corticosteroids >20 mg/day, prednisone or equivalent
* Clinical conditions requiring treatment with oral or parenteral anticoagulants or antiplatelet agents unless treatment can be discontinued 7 days (or 5 half-lives) prior to initiation of study treatment (except used as flushes for indwelling catheters)
* History of severe allergic or anaphylactic reaction to humanized or murine monoclonal antibodies
* Known hypersensitivity or allergy to murine products or any component of the obinutuzumab, rituximab, idasanutlin, or venetoclax formulation
* Current or history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection: positive for hepatitis B surface antigen (HBsAg), total hepatitis B core antibody (HBcAb), or HCV antibody at screening
* History of progressive multifocal leukoencephalopathy (PML)
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Evidence of any significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results
* Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by study treatment, such as severe hereditary coagulation disorders or insulin-dependent diabetes mellitus that is not optimally controlled with medical management (example, presence of ketoacidosis)
* Major surgical procedure other than for diagnosis within 28 days prior to Day 1 of Cycle 1, or anticipation of a major surgical procedure during the study
* Inadequate hematologic function (unless due to underlying lymphoma), defined as follows: Hemoglobin less than (<) 9 grams per decilitre (g/dL), absolute neutrophil count (ANC) <1.5*10^9 cells per liter (cells/L), platelet count <75*10^9 cells/L
* Any of the following abnormal laboratory values (unless due to underlying lymphoma): International normalized ratio (INR) or prothrombin time (PT) >1.5*upper limit of normal (ULN) in the absence of therapeutic anticoagulation; partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) >1.5*ULN in the absence of a lupus anticoagulant
* Life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- United States (7):
  - University of Colorado, Aurora, Colorado
  - The University of Chicago Medical Center, Chicago, Illinois
  - Norton Cancer Institute - Dutchmans, Louisville, Kentucky
  - Mount Sinai Medical Center, New York, New York
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - Swedish Cancer Inst., Seattle, Washington
- Australia (3):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Germany (5):
  - Klinikum Augsburg, Augsburg
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Klinikum rechts der Isar der TU München, München
  - Universitätsklinikum Würzburg; Studienzentrale Hämatologie/Onkologie, Würzburg
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Auckland Clinical Studies Limited, Grafton
- South Korea (4):
  - Keimyung University Dongsan Medical Center, Daegu
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 Participants (ITT population) were enrolled at 13 sites in the USA, Australia, South Korea, New Zealand and Germany during the dose escalation phase. 1 participant was undefined as the diagnosis at study entry was not provided.
  Due to the study's pre-mature termination, the planned Dose Expansion Phase did not take place for both arms DLBCL and FL.
Pre-assignment Details: The study was prematurely terminated because of the overall modest benefit achieved with MTD during the escalation phase.
  In each DLBCL and FL arm, participants are in Safety Cohort, Cohort 1, Cohort 2, Cohort 3 and Cohort 3- Not defined (DLBCL only).
  All Adverse Events are reported per Cohort rather than per Arm.
Groups:
- Dose Escalation DLBCL and FL Safety Cohort; Dose Escalation DLBCL and FL Cohort 1: Idasanutlin 100 mg + Venetoclax 200 mg + Obinutuzumab 1000 mg
- Dose Escalation DLBCL and FL Cohort 2: Idasanutlin 150 mg + Venetoclax 200 mg + Obinutuzumab 1000 mg
- Dose Escalation DLBCL and FL Cohort 3: Idasanutlin 100 mg + Venetoclax 400 mg + Obinutuzumab 1000 mg
- Not Defined for DLBCL or FL Subgroups Cohort 3: Idasanutlin 100 mg+ Venetoclax 200mg + obinutuzumab 1000 mg
Period: Overall Study
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escalation DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Started | 9 | 6 | 7 | 6 | 1
Completed | 0 (The study was terminated after escalation phase. The planned expansion phase did not take place due to the early termination.) | 0 (The study was terminated after escalation phase. The planned expansion phase did not take place due to the early termination.) | 0 (The study was terminated after escalation phase. The planned expansion phase did not take place due to the early termination.) | 0 (The study was terminated after escalation phase. The planned expansion phase did not take place due to the early termination.) | 0 (The study was terminated after escalation phase. The planned expansion phase did not take place due to the early termination.)
Not Completed | 9 | 6 | 7 | 6 | 1
Not completed — discontinued due to worsening of pre-existing medical condition | 1 | 0 | 0 | 0 | 0
Not completed — Progression of disease | 0 | 0 | 0 | 1 | 0
Not completed — Death | 6 | 2 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1
Not completed — Study terminated by sponsor | 2 | 4 | 4 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose-Escalation DLBCL and FL Safety Cohort; Dose-Escalation DLBCL and FL Cohort 1: Idasanutlin 100 mg + venetoclax 200 mg + obinutuzumab 1000 mg
- Dose Escaltion DLBCL and FL Cohort 2: Idasanutlin 150 mg + venetoclax 200 mg + obinutuzumab 1000 mg
- Total: Total of all reporting groups
Arm/Group | Dose-Escalation DLBCL and FL Safety Cohort | Dose-Escalation DLBCL and FL Cohort 1 | Dose Escaltion DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3 | Total
Number analyzed (Participants) | 9 | 6 | 7 | 6 | 1 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: ITT
  Years | 58.6 (15.5) | 68.5 (8.7) | 72.4 (8.6) | 74.3 (5.5) | 25.0 (0) | 66.1 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    Female | 3 | 3 | 3 | 3 | 0 | 12
    Male | 6 | 3 | 4 | 3 | 1 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 6 | 7 | 6 | 1 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 7 | 5 | 6 | 2 | 1 | 21
  More than one race | 0 | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: RP2D of Idasanutlin When Given in Combination With Obinutuzumab or Rituximab
Description: It was planned to be identified in escalation and carried over in expansion phases. However the expansion phase did not take place. phases.
  The study was closed because at escalation doses 100 (in combination with venetoclax 400 mg) and 150 mg (in combination with venetoclax 200 mg) Idasanutlin, the benefit was mild. The study was terminated at the escalation phase with DLTs showing AEs in all cohorts. The subpopulations of DLBCL and FL were showed no difference in their genetic subtype make-up, therefore, Cohorts Safety, 1, 2, 3 contain both populations.
  The safety cohort had a different venetoclax schedule of 5 days to ensure safety. Remaining cohorts used a 10 days schedule. No RP2D was identified in the Cohorts 1 and 3.
Time Frame: Cycle 1 Day 1 up to Cycle 2 Day 28 (each cycle = 28 days)
Population: Safety Population
Measure: Number; unit: mg
Groups:
- Dose Escaltion DLBCL and FL Cohort 1: Idasanutlin 100 mg + venetoclax 200 mg + obinutuzumab 1000 mg
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escaltion DLBCL and FL Cohort 1 | Dose Escaltion DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 9 | 6 | 7 | 6 | 1
mg | NA — No qualifying value data available | NA — No qualifying value data available | 150 | NA — No qualifying value data available | NA — No qualifying value data available

2. Primary Outcome: RP2D of Venetoclax When Given in Combination With Obinutuzumab or Rituximab
Description: It was planned to be identified in escalation and carried over in expansion phases. However the expansion phase did not take place.
  The study was closed because at escalation doses 200 (in combination with 150 mg idasanutlin) and 400 (in combination with 100 mg idasanutlin) mg Venetoclax, the benefit was mild. The study was terminated at the escalation phase with DLTs showing AEs in all cohorts.
  The safety cohort had a different venetoclax schedule of 5 days to ensure safety. Remaining cohorts used a 10 days schedule. No RP2D was identified in the Cohorts 1 and 3.
Time Frame: Cycle 1 Day 1 up to Cycle 2 Day 28 (each cycle = 28 days)
Population: Safety Population
Measure: Number; unit: mg
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escaltion DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 9 | 6 | 7 | 6 | 1
mg | NA — No qualifying value data available | NA — No qualifying value data available | 200 | NA — No qualifying value data available | NA — No qualifying value data available

3. Primary Outcome: Percentage of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT is defined as any one of the following events occurring during first two Cycles of treatment and assessed by the investigator as clearly not related to patient's underlying disease: - Any Grade 5 adverse event (AE) unless unequivocally due to the underlying malignancy or extraneous causes; - AE of any grade that leads to a delay of more than 14 days at the start of next treatment cycle; - Hematologic AEs (neutropenia, thrombocytopenia); - Non-hematologic AE, except IRRs, laboratory TLS without manifestations of clinical TLS, AST or ALT, diarrhea, nausea or vomiting, fatigue, asthenia, anorexia, or constipation, hepatic transaminase.
Time Frame: Cycle 1 Day 1 up to Cycle 2 Day 28 (each cycle = 28 days)
Population: Safety-Evaluable Patients
Measure: Number; unit: Percentage of Participants
Groups:
- Dose Escaltion DLBCL and FL Safety Cohort; Dose Escaltion DLBCL and FL Cohort 1: Idasanutlin 100 mg + venetoclax 200 mg + obinutuzumab 1000 mg
Arm/Group | Dose Escaltion DLBCL and FL Safety Cohort | Dose Escaltion DLBCL and FL Cohort 1 | Dose Escaltion DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 9 | 6 | 7 | 6 | 1
Percentage of Participants | 0 | 16.7 | 28.6 | 16.7 | 0

4. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a casual relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporarily associated with the use of pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: From Baseline up to approximately 48 months
Population: Safety Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Dose Escaltion DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escalation DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 9 | 6 | 7 | 6 | 1
Percentage of Participants | 100 | 100 | 100 | 100 | 0

5. Primary Outcome: Percentage of Participants With Complete Response (CR), Determined by an Independent Review Committee (IRC) on the Basis of Positron Emission Tomography-Computed Tomography (PET-CT) Scans Using Modified Lugano 2014 Criteria
Description: The study plan was for the IRC to analyze the efficacy results in participants from the expansion phase (Part II), but the expansion phase was not opened (i.e., no enrollment) because the sponsor decided to terminate the study early due to the modest benefit achieved with the maximum tolerated dose during the dose escalation phase (Part I). Therefore the result data not derived and not reported.
Time Frame: At end of Induction (EOI) (within 6 to 8 weeks after Cycle 6 Day 1 [up to approximately 28 weeks] [each cycle = 28 days])
Population: The study plan was for the IRC to analyze the efficacy results in participants from the expansion phase (Part II), but the expansion phase was not opened (i.e., no enrollment) because the sponsor decided to terminate the study early due to the modest benefit achieved with the maximum tolerated dose during the dose escalation phase (Part I).
Arm/Group | Dose-Escalation DLBCL and FL Safety Cohort | Dose-Escalation DLBCL and FL Cohort 1 | Dose Escaltion DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With CR, Determined by the Investigator on the Basis of PET-CT Scans Using Modified Lugano 2014 Criteria
Description: The investigator evaluated responses at the end of induction treatment using Lugano 2014 criteria for malignant lymphoma for a PET-CT based complete response (CR), which required a complete metabolic response with a score of 1, 2 or 3 with or without a residual mass in lymph nodes and extralymphatic sites on the PET 5-point scale for 18-fluorodeoxyglucose (FDG) uptake (1 = no uptake above background; 2 = uptake less than or equal to [<=] mediastinum; 3 = uptake greater than [>] mediastinum and <= liver; 4 = uptake moderately > liver; 5 = uptake markedly > liver and/or new lesions). The CR criteria were slightly modified to require normal bone marrow by morphology (if intermediate, immunohistochemistry negative). PET-CT scans were performed at end of induction only on participants who had received at least 2 cycles of induction treatment; those without a post-baseline tumor assessment were considered non-responders.
Time Frame: At EOI (6 to 8 weeks after Cycle 6 Day 1 [up to approximately 28 weeks] [each cycle = 28 days]
Population: ITT Population; exploratory analysis of the dose escalation phase (Part I). The study plan was for efficacy analyses to be based on responses in participants enrolled during the expansion phase (Part II), but it was not opened (i.e., no enrollment) and at the study was terminated early.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Groups:
- Dose Escalation DLBCL and FL Cohort 2: Idasanutlin 150 mg + venetoclax 400 mg + obinutuzumab 1000 mg
Arm/Group | Dose Escaltion DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escalation DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 9 | 6 | 7 | 6 | 1
Percentage of Participants | 22.2 [4.10 to 54.96] | 16.7 [0.85 to 58.18] | 28.6 [5.34 to 65.87] | 16.7 [0.85 to 58.18] | 0 [0.00 to 95.00]

7. Secondary Outcome: Percentage of Participants With CR, Determined by the IRC on the Basis of CT Scans Alone Using Modified Lugano 2014 Criteria
Description: The IRC was to evaluate responses at the end of induction treatment using the Lugano 2014 response criteria for malignant lymphoma for a computed tomography (CT)-based complete response (CR). The CR criteria required to complete radiologic response with all of the following: target nodal masses must regress to less than or equal to 1.5 centimeters in the longest transverse diameter of a lesion [LDi]; no extralymphatic sites of disease; no non-measured or new lesions; enlarged organs regressing to normal size; and bone marrow normal by morphology (if indeterminate, immunochemistry negative). CT scans were performed at end of induction only on participants who had received at least 2 cycles of induction treatment; those without a post-baseline tumor assessment were to be considered non-responders. Therefore the result data not derived and not reported.
Time Frame: At EOI (6 to 8 weeks after Cycle 6 Day 1 [up to approximately 28 weeks] [each cycle = 28 days]
Population: The study plan was for the IRC to analyze the efficacy results in participants from the expansion phase (Part II), but the expansion phase was not opened (i.e. , no enrollment) because the sponsor decided to terminate the study early due to the modest benefit achieved with the maximum tolerated dose during the dose escalation phase (Part I).
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escaltion DLBCL and FL Cohort 1 | Dose Escaltion DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants With CR, Determined by the Investigator on the Basis of CT Scans Alone Using Modified Lugano 2014 Criteria
Description: The investigator evaluated responses at the end of induction treatment using the Lugano 2014 response criteria for malignant lymphoma for a computed tomography (CT)-based complete response (CR). The CR criteria required a complete radiologic response with all of the following: target nodes/nodal masses must regress to less than or equal to 1.5 centimeters in the longest transverse diameter of a lesion (LDi); no extralymphatic sites of disease; no non-measured or new lesions; enlarged organs regressing to normal size; and bone marrow normal by morphology (if indeterminate, immunohistochemistry negative). CT scans were performed at end of induction only on participants who received at least 2 cycles of Induction treatment; those without a post-baseline tumor assessment were to be considered non-responders. This outcome measure therefore not derived and not reported.
Time Frame: At EOI (6 to 8 weeks after Cycle 6 Day 1 [up to approximately 28 weeks] [each cycle = 28 days]
Population: ITT Population; exploratory analysis of the dose escalation phase (Part I). The study plan was for efficacy analyses to be based on responses in participants enrolled during expansion phase (Part II), but it was not opened (i.e., no enrollment) and at the study was terminated early.
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escalation DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants With Objective Response, Determined by the IRC on the Basis of PET-CT Scans Using Modified Lugano 2014 Criteria
Description: The IRC was to evaluate responses at the end of induction treatment using Luagno 2014 criteria for malignant lymphoma for a PET-CT based objective response: either a complete (CR) or partial response (PR). A CR required a complete metabolic response with a score of 1, 2 or 3 on the PET 5-point scale (5PS) for 18-fluorodeoxyglucose (FDG) uptake (scores range from 1 [no uptake above background] to 5 [uptake markedly higher than liver and/or new lesions]), with or without a residual mass in lymph nodes and extralymphatic sites; and a PR required a partial metabolic response with a score 4 or 5 on the 5PS with reduced 18-FDG uptake compared with baseline and residual mass(es) of any size. For bone marrow involvement, the CR criteria required no evidence of FDG-avid disease, and the PR criteria required residual uptake higher than in normal marrow but reduced compared with baseline. Therefore the result data not derived and not reported. The study was pre-maturely terminated.
Time Frame: At EOI (6 to 8 weeks after Cycle 6 Day 1 [up to approximately 28 weeks] [each cycle = 28 days]
Population: The study plan was for the IRC to analyze the efficacy results in participants from the expansion phase (Part II)., but the expansion phase was not opened (i.e., no enrollment) because the sponsor decided to terminate the study early due to the modest benefit achieved with the maximum tolerated dose during the dose escalation phase (Part I).
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escaltion DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With Objective Response, Determined by the Investigator on the Basis of PET-CT Scans Using Modified Lugano 2014 Criteria
Description: The investigator was to evaluate responses at end of induction treatment using Lugano 2014 criteria for malignant lymphoma for a PET-CT based objective response: either a complete (CR) or partial response (PR). A CR required a complete metabolic response with a score of 1, 2, or 3 on the PET 5-point scale (5PS) for 18-fluorodeoxyglucose (FDG) uptake (scores range from 1 [no uptake above background] to 5 [uptake markedly higher than liver and/or new lesions]), with or without a residual mass in lymph nodes and extralymphatic sites; and a PR required a partial metabolic response with a score of 4 or 5 on the 5PS with reduced 18-FDG uptake compared with baseline and residual mass(es) of any size. For bone marrow involvement, the CR criteria required no evidence of FDG-avid disease, and the PR criteria required residual uptake higher than in normal marrow but reduced compared with baseline. Participants without a post-baseline tumor assessment were to be considered non-responders.
Time Frame: At EOI (6 to 8 weeks after Cycle 6 Day 1 [up to approximately 28 weeks] [each cycle = 28 days]
Population: ITT Population
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escalation DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 9 | 6 | 7 | 6 | 1
Percentage of Participants | 33.3 [9.77 to 65.51] | 16.7 [0.85 to 58.18] | 28.6 [5.34 to 65.87] | 33.3 [6.28 to 72.87] | 0 [0.00 to 95.00]

11. Secondary Outcome: Percentage of Participants With Objective Response, Determined by the IRC on the Basis of CT Scans Alone Using Modified Lugano 2014 Criteria
Description: The IRC was to evaluate responses at the end of induction treatment using the Lugano 2014 response criteria for malignant lymphoma for a CT-based objective response: either a complete (CR) or partial response (PR). The CR criteria required a complete radiologic response with all of the following: target nodes/nodal masses must regress to less than or equal to 1.5 cm in the LDi; no extralymphatic sites of disease; no non-measured or new lesions; enlarged organs regressing to normal size; and bone marrow normal by morphology (if indeterminate, immunohistochemistry negative). The PR criteria required all of the following: a >=50% decrease in sum of the product of perpendicular diameters of up to 6 target measurable nodes and extranodal sites; no new lesions; non-measured lesion that is absent/nomal, regressed, but no increase; and spleen must have regressed by >50% in length. Therefore the result data not derived and not reported. The study was pre-maturely terminated.
Time Frame: At EOI (6 to 8 weeks after Cycle 6 Day 1 [up to approximately 28 weeks] [each cycle = 28 days]
Population: as for outcome 9
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escalation DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants With Objective Response at EOI, Determined by the Investigator on the Basis of CT Scans Alone Using Modified Lugano 2014 Criteria
Description: The investigator was to evaluate responses at the end of induction treatment using Lugano 2014 response criteria for malignant lymphoma for a CT-based objective response: either a complete (CR) or partial response (PR). The CR criteria required a complete radiologic response with all of the following: target nodes/nodal masses must regress to less than or equal to 1.5 cm in LDi; no extralymphatic sites of disease; no non-measured or new lesions; enlarged organs regressing to normal size; and bone marrow normal by morphology (if indeterminate, immunohistochemistry negative). The PR criteria required all of the following: a >=50% decrease in sum of the product of perpendicular diameters up to 6 target measurable nodes and extranodal sites; no new lesions; non-measured lesion that is absent/normal, regressed, but no increase; and spleen must have regressed by >50% in length. The study was pre-maturely terminated at escalation phase.
Time Frame: At EOI (6 to 8 weeks after Cycle 6 Day 1 [up to approximately 28 weeks] [each cycle = 28 days]
Population: as for outcome 9
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escalation DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants With Objective Response During the Study, Determined by the Investigator on the Basis of CT Scans Alone Using Modified Lugano 2014 Criteria
Description: as for outcome 12
Time Frame: From Day 1 of Cycle 1 (cycle length = 28 days) up to approximately 48 months
Population: as for outcome 9
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escalation DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Observed Serum Concentration of Obinutuzumab in Participants With FL
Description: Observed Serum Concentration of Obinutuzumab in Participants With FL was planned to be determined as part of the pharmacokinetics analyses during the expansion phase which did not take place.
  The study was prematurely terminated because of the overall modest benefit achieved with MTD during the escalation phase (Part 1); Phase II of the study (expansion) was never initiated. No result data was derived, therefore no result was reported.
  The result data not derived due to early termination of the study by the sponsor's decision and did not reach the end of study.
Time Frame: From Day 1 of Cycle 1 (cycle length = 28 days) up to approximately 48 months (detailed timeframe is mentioned in outcome measure description)
Population: ITT Population was planned. Due to the pre-mature study termination, no participants were available for this endpoint and result data were not collected.
Groups:
- Dose Escalation FL Safety Cohort; Dose Escalation FL Cohort 1: Idasanutlin 100 mg + venetoclax 200 mg + obinutuzumab 1000 mg
- Dose Escalation FL Cohort 2: Idasanutlin 150 mg + venetoclax 200 mg + obinutuzumab 1000 mg
- Dose Escalation FL Cohort 3: Idasanutlin 100 mg + venetoclax 400 mg + obinutuzumab 1000 mg
Arm/Group | Dose Escalation FL Safety Cohort | Dose Escalation FL Cohort 1 | Dose Escalation FL Cohort 2 | Dose Escalation FL Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Observed Serum Concentration of Obinutuzumab in Participants With DLBCL
Description: Observed Serum Concentration of Obinutuzumab in Participants With DLBCL was planned to be determined as part of the pharmacokinetics analyses during the expansion phase which did not take place.
  The study was prematurely terminated because of the overall modest benefit achieved with MTD during the escalation phase (Part 1); Phase II of the study (expansion) was never initiated. No result data was derived, therefore no result was reported.
Time Frame: Induction: Pre-dose (any time prior to dose on same day) and 30 min post-dose on Day 1 of Cycle 1; Pre-dose (within 5 hrs prior to dose) and 30 min post-dose on Day 1 of Cycles 2, 4 and 6 (each cycle = 28 days)
Population: as for outcome 14
Groups:
- Dose Escalation DLBCL Safety Cohort 2; Dose Escalation DLBCL Cohort 1: Idasanutlin 100 mg + venetoclax 200 mg + obinutuzumab 1000 mg
- Dose Escaltion DLBCL Cohort 2: Idasanutlin 150 mg + venetoclax 200 mg + obinutuzumab 1000 mg
- Dose Escalation DLBCL Cohort 3: Idasanutlin 100 mg + venetoclax 400 mg + obinutuzumab 1000 mg
Arm/Group | Dose Escalation DLBCL Safety Cohort 2 | Dose Escalation DLBCL Cohort 1 | Dose Escaltion DLBCL Cohort 2 | Dose Escalation DLBCL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Observed Serum Concentration of Rituximab in Participants With FL
Description: Observed Serum Concentration of Rituximab in Participants With FL was planned to be determined as part of the pharmacokinetics analyses during the expansion phase which did not take place.
  The study was prematurely terminated because of the overall modest benefit achieved with MTD during the escalation phase (Part 1); Phase II of the study (expansion) was never initiated. No result data was derived, therefore no result was reported.
Time Frame: Induction: Pre-dose (any time prior to dose on same day) on Day 1 of Cycle 1; Pre-dose (within 5 hrs prior to dose) on Day 1 of Cycles 2, 4, 6; 30 min post-dose on Day 1 of Cycles 1 and 6 (each cycle = 28 days)
Population: as for outcome 14
Arm/Group | Dose Escalation FL Safety Cohort | Dose Escalation FL Cohort 1 | Dose Escalation FL Cohort 2 | Dose Escalation FL Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Observed Serum Concentration of Rituximab in Participants With DLBCL
Description: Observed Serum Concentration of Rituximab in Participants With DLBCL was planned to be determined as part of the pharmacokinetics analyses during the expansion phase which did not take place.
  The study was prematurely terminated because of the overall modest benefit achieved with MTD during the escalation phase (Part 1); Phase II of the study (expansion) was never initiated. No result data was derived, therefore no result was reported.
Time Frame: as for outcome 14
Population: as for outcome 14
Groups:
- Dose Escaltion DLBCL Safety Cohort; Dose Escalation DLBCL Cohort 1: Idasanutlin 100 mg + venetoclax 200 mg + obinutuzumab 1000 mg
Arm/Group | Dose Escaltion DLBCL Safety Cohort | Dose Escalation DLBCL Cohort 1 | Dose Escaltion DLBCL Cohort 2 | Dose Escalation DLBCL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Observed Plasma Concentration of Idasanutlin in Participants With FL
Description: Observed Plasma Concentration of Idasanutlin in Participants With FL was planned to be determined as part of the pharmacokinetics analyses during the expansion phase which did not take place.
  The study was prematurely terminated because of the overall modest benefit achieved with MTD during the escalation phase (Part 1); Phase II of the study (expansion) was never initiated. No result data was derived therefore no result was reported
Time Frame: From Day 1 of Cycle 1 up to Day 5 of Cycle 4 (each cycle = 28 days) (detailed timeframe is mentioned in outcome measure description)
Population: as for outcome 14
Arm/Group | Dose Escalation FL Safety Cohort | Dose Escalation FL Cohort 1 | Dose Escalation FL Cohort 2 | Dose Escalation FL Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Secondary Outcome: Observed Plasma Concentration of Idasanutlin in Participants With DLBCL
Description: Observed Plasma Concentration of Idasanutlin in Participants With DLBCL was planned to be determined as part of the pharmacokinetics analyses during the expansion phase which did not take place.
  The study was prematurely terminated because of the overall modest benefit achieved with MTD during the escalation phase (Part 1); Phase II of the study (expansion) was never initiated. No result data was derived therefore no result was reported
Time Frame: as for outcome 18
Population: as for outcome 14
Groups:
- Dose Escalation DLBCL Safety Cohort; Dose Escalation DLBCL Cohort 1: Idasanutlin 100 mg + venetoclax 200 mg + obinutuzumab 1000 mg
Arm/Group | Dose Escalation DLBCL Safety Cohort | Dose Escalation DLBCL Cohort 1 | Dose Escaltion DLBCL Cohort 2 | Dose Escalation DLBCL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Observed Plasma Concentration of Venetoclax in Participants With FL
Description: Observed Plasma Concentration of Venetoclax in Participants With FL was planned to be determined as part of the pharmacokinetics analyses during the expansion phase which did not take place.
  The study was prematurely terminated because of the overall modest benefit achieved with MTD during the escalation phase (Part 1); Phase II of the study (expansion) was never initiated.
Time Frame: as for outcome 18
Population: as for outcome 14
Arm/Group | Dose Escalation FL Safety Cohort | Dose Escalation FL Cohort 1 | Dose Escalation FL Cohort 2 | Dose Escalation FL Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Secondary Outcome: Observed Plasma Concentration of Venetoclax in Participants With DLBCL
Description: Observed Plasma Concentration of Venetoclax in Participants With DLBCL was planned to be determined as part of the pharmacokinetics analyses during the expansion phase which did not take place.
  The study was prematurely terminated because of the overall modest benefit achieved with MTD during the escalation phase (Part 1); Phase II of the study (expansion) was never initiated.
Time Frame: as for outcome 18
Population: as for outcome 14
Groups:
- Dose Escaltion DLBCL Cohort 1: Idasanutlin 100 mg + venetoclax 200 mg + obinutuzumab 1000 mg
- Dose Escalation DLBCL Cohort 2: Idasanutlin 150 mg + venetoclax 200 mg + obinutuzumab 1000 mg
Arm/Group | Dose Escaltion DLBCL Safety Cohort | Dose Escaltion DLBCL Cohort 1 | Dose Escalation DLBCL Cohort 2 | Dose Escalation DLBCL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline Up to Approximately 3 Years
Description: Reported: Safety Population. During the Safety Follow-up Period, non-Serious Adverse Events occurred at the 5% frequency threshold. There was no non-SAEs occurred reported in Dose Escalation DLBCL only Cohort 3 Not Defined arm.
Arm/Group | Dose Escalation DLBCL and FL Safety Cohort | Dose Escalation DLBCL and FL Cohort 1 | Dose Escalation DLBCL and FL Cohort 2 | Dose Escalation DLBCL and FL Cohort 3 | Not Defined for DLBCL or FL Subgroups Cohort 3
All-Cause Mortality (participants affected / at risk) | 6/9 | 2/6 | 2/7 | 2/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/9 | 3/6 | 4/7 | 4/6 | 0/1
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6 | 7/7 | 6/6 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation DLBCL and FL Safety Cohort (N=9) | Dose Escalation DLBCL and FL Cohort 1 (N=6) | Dose Escalation DLBCL and FL Cohort 2 (N=7) | Dose Escalation DLBCL and FL Cohort 3 (N=6) | Not Defined for DLBCL or FL Subgroups Cohort 3 (N=1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation DLBCL and FL Safety Cohort (N=9) | Dose Escalation DLBCL and FL Cohort 1 (N=6) | Dose Escalation DLBCL and FL Cohort 2 (N=7) | Dose Escalation DLBCL and FL Cohort 3 (N=6) | Not Defined for DLBCL or FL Subgroups Cohort 3 (N=1)
ANAEMIA (Blood and lymphatic system disorders) | 4 (5) | 1 (1) | 4 (4) | 3 (6) | NA
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 3 (8) | 1 (1) | NA
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | NA
NEUTROPENIA (Blood and lymphatic system disorders) | 7 (13) | 5 (8) | 7 (20) | 5 (21) | NA
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 7 (9) | 4 (5) | 7 (13) | 5 (6) | NA
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | NA
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
EYE DISORDER (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
EYE PAIN (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
PHOTOPHOBIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
VISION BLURRED (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | NA
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | NA
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | NA
DIARRHOEA (Gastrointestinal disorders) | 5 (9) | 3 (3) | 4 (6) | 4 (10) | NA
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | NA
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | NA
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
NAUSEA (Gastrointestinal disorders) | 6 (14) | 4 (6) | 3 (3) | 3 (8) | NA
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
TONGUE HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | NA
VOMITING (Gastrointestinal disorders) | 3 (5) | 3 (3) | 1 (1) | 2 (2) | NA
CHEST PAIN (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | NA
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | NA
FATIGUE (General disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | NA
NON-CARDIAC CHEST PAIN (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | NA
OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
UNEVALUABLE EVENT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | NA
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
MUCOSAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | NA
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | NA
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | NA
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | NA
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | NA
MEDICATION ERROR (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
PRODUCT ADMINISTRATION ERROR (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
PRODUCT DOSE OMISSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
WRONG TECHNIQUE IN PRODUCT USAGE PROCESS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
ALANINE AMINOTRANSFERASE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | NA
AMYLASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | NA
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | NA
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | NA
PLATELET COUNT DECREASED (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | NA
RESPIROVIRUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
SERUM FERRITIN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (4) | 0 (0) | 1 (5) | 2 (7) | NA
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | NA
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | NA
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | NA
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
HYPOPHAGIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | NA
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | NA
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | NA
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | NA
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | NA
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
DIZZINESS (Nervous system disorders) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | NA
HEADACHE (Nervous system disorders) | 3 (5) | 1 (2) | 2 (2) | 1 (1) | NA
NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
PARAESTHESIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
RADICULAR PAIN (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
DYSURIA (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | NA
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | NA
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
LOWER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | NA
ERYTHEMA AB IGNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | NA
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | NA
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
FLUSHING (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
LYMPHATIC FISTULA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
Dose expansion part of the study did not take place. AEs were not differentiated for DLBCL and FL arms since these are sub mutations of disease which does nor show differences in AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT03135262/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT03135262/SAP_001.pdf